CLINICAL TRIAL: NCT01696552
Title: Patient-specific Positioning Guides (PSPG) Technique Versus Conventional Technique in Total Knee Arthroplasty - a Prospective Randomized Study.
Brief Title: Patient-specific Positioning Guides (PSPG) Technique Versus Conventional Technique in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Betanien Hospital (Other); Sykehuset Telemark (Other Government); Vestre Viken Hospital Trust (Other)
Responsible Party: Principal Investigator, Stephan M Rohrl, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011/7613; 2010/2056 (Other: Regional Committee for Medical Health Research Ethics West)
Record Dates: First submitted 2012-08-19; First posted 2012-10-01 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Gonarthritis
Keywords: Gonarthritis; TKR; Conventional; Positioning Guides; PSPG; CT Perth
MeSH Terms: interventions — tokaratoxin 2; Cimetidine; Amino Acid Motifs

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TKR with Positioning Guides (PSPG) (Active Comparator): Use of PSPG (Signature, Materialise) in TKR (Vanguard Total Knee System, Biomet)
  Interventions: Procedure: TKR with Positioning Guides (PSPG)
- TKR with Conventional Technique (Active Comparator): TKR (Vanguard Total Knee System, Biomet), Conventional Technique
  Interventions: Procedure: TKR with Conventional Technique

INTERVENTIONS:
Procedure: TKR with Positioning Guides (PSPG) — TKR (Vanguard Total Knee System, Biomet) with PSPG (Signature, Materialise) technique
  Other Names: Vanguard Total Knee System, Biomet; Signature, Materialise
  Arms: TKR with Positioning Guides (PSPG)
Procedure: TKR with Conventional Technique — TKR (Vanguard Total Knee System, Biomet) with Conventional Technique
  Other Names: Vanguard Total Knee System, Biomet
  Arms: TKR with Conventional Technique

SUMMARY:
A Prospective, randomized, clinical controlled study comparing conventional knee arthroplasty and the Patient-specific positioning guides (PSPG) (Signature Patient Care, Materialise) using the Vanguard Total Knee System (Biomet)

DETAILED DESCRIPTION:
Background: Use of PSPG in TKR is a relative new technique and already widely used. PSPG, based on MRI data, fit directly into the patient's anatomy and enable total knee replacement without use of traditional invasive instrumentation. Data showing extra benefit of this technique compared to conventional TKR technique are not widely available.

Aim: To determine the safety of this new surgical technique compared to conventional TKR and whether a clinical, functional and financial benefit can be achieved.

Methods: 200 patients with primary osteoarthritis will be randomized to 2 groups. 30 patients in each group will be included in the RSA section of the study. Participating hospitals UOS Ullevål, Vestre Viken, Sykehuset Telemark and Betanien Hospital Skien. Inclusion started Aug. 2011. Clinical scoring: KSS, KOOS, EQ-5D and VAS will be examined at inclusion, after 3 months, and at the 1 and 2 year control. RSA before discharge on day 2, 3 months, 1 year, 2 years. RSA images will be sent blinded to CIRRO (Center for Implant and Radiostereometric Research Oslo Orthopaedic Centre, Oslo University Hospital) for image analysis. Standing HKA: preoperatively and after 3 months. X-ray will be taken pre-operatively, postoperative day 3, after 3 months and after 5 and 10 years. CT Perth after 3 months for measuring alignment. A cost-benefit analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Man and women elder than 18 years old with knee osteoarthritis
2. Informed consent

Exclusion Criteria:

1. Active infection.
2. Under 50 years.
3. Revision arthroplasty.
4. Marked bone loss which could preclude adequate fixation of the device.
5. Non-cooperative subjects.
6. Parkinson's Disease or other neurologic and muscular disorders
7. Severe vascular insufficiency of the affected limb.
8. Severe instability or deformity of the ligaments and / or surrounding soft tissue which may preclude stability of the device.
9. Paget's disease
10. Rheumatoid Arthritis and other systemic diseases
11. Patients with rigid hip joints
12. Known metal allergy
13. Patients can only join the study with 1 operated knee arthroplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-01 (Actual); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Assessing total knee implant positioning using PSPG compared with the conventional method in TKR | 3 months
  Measurement of knee implant positioning by using the CT Perth protocol

SECONDARY OUTCOMES:
Clinical Functional Result | 2 yrs
  KOOS (Knee injury and Osteoarthritis Outcome Score), American knee society score, EQ-5D and pain score (NRS) will be registered pre-operatively, after 3 months and after 1 and 2 years. Scores of the 2 groups will be compared.
Operating Time | 1 day
Component Stability | 2 yrs
  RSA
Cost to Benefit from a Health Economic Perspective | 1 year
  Cost-benefit analysis
X-ray analysis | 10 yrs
  Standing HKA (Hip, Knee, Ankle-long axis images): preoperatively and after 3 months. If there is a extension deficit a X-HKA will be performed 12 months postoperatively.
  X-ray front, side and patella 'sky view' will be taken pre-operatively, postoperative day 3, after 5 and 10 years. Alignment and possible osteolytic development will be recorded in both groups.
Perioperative Morbidity | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Stephan M Röhrl, MD, PhD, Principal Investigator — Oslo Univerity Hospital, Oslo, Norway; Justin van Leeuwen, MD, Principal Investigator — Betanien Hospital Skien, Skien, Norway; Bjarne Grøgaard, MD, PhD, Principal Investigator — Oslo University Hospital, Oslo, Norway; Finnur Snorrason, MD, PhD, Principal Investigator — Vestre Viken HF, Drammen Hospital, Drammen, Norway; Hilde Apold, MD, PhD, Principal Investigator — Sykehuset Telemark
Locations (4):
- Norway (4):
  - Vestre Viken HF, Drammen, Buskerud
  - Center for Implant and Radiostereometric Research Oslo, Oslo University Hospital, Oslo, Olso
  - Sykehuset Telemark, Skien, Telemark
  - Betanien Hospital Skien, Skien, Telemark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Valstar ER, Gill R, Ryd L, Flivik G, Borlin N, Karrholm J. Guidelines for standardization of radiostereometry (RSA) of implants. Acta Orthop. 2005 Aug;76(4):563-72. doi: 10.1080/17453670510041574. PMID 16195075
- [Background] Ritter MA, Faris PM, Keating EM, Meding JB. Postoperative alignment of total knee replacement. Its effect on survival. Clin Orthop Relat Res. 1994 Feb;(299):153-6. PMID 8119010
- [Background] Chauhan SK, Clark GW, Lloyd S, Scott RG, Breidahl W, Sikorski JM. Computer-assisted total knee replacement. A controlled cadaver study using a multi-parameter quantitative CT assessment of alignment (the Perth CT Protocol). J Bone Joint Surg Br. 2004 Aug;86(6):818-23. doi: 10.1302/0301-620x.86b6.15456. PMID 15330021
- [Background] Klatt BA, Goyal N, Austin MS, Hozack WJ. Custom-fit total knee arthroplasty (OtisKnee) results in malalignment. J Arthroplasty. 2008 Jan;23(1):26-9. doi: 10.1016/j.arth.2007.10.001. PMID 18165024
- [Background] Fehring TK, Odum S, Griffin WL, Mason JB, Nadaud M. Early failures in total knee arthroplasty. Clin Orthop Relat Res. 2001 Nov;(392):315-8. doi: 10.1097/00003086-200111000-00041. PMID 11716402
- [Background] Ng VY, DeClaire JH, Berend KR, Gulick BC, Lombardi AV Jr. Improved accuracy of alignment with patient-specific positioning guides compared with manual instrumentation in TKA. Clin Orthop Relat Res. 2012 Jan;470(1):99-107. doi: 10.1007/s11999-011-1996-6. PMID 21809150
- [Background] Karrholm J, Borssen B, Lowenhielm G, Snorrason F. Does early micromotion of femoral stem prostheses matter? 4-7-year stereoradiographic follow-up of 84 cemented prostheses. J Bone Joint Surg Br. 1994 Nov;76(6):912-7. PMID 7983118
- [Background] Ryd L, Albrektsson BE, Carlsson L, Dansgard F, Herberts P, Lindstrand A, Regner L, Toksvig-Larsen S. Roentgen stereophotogrammetric analysis as a predictor of mechanical loosening of knee prostheses. J Bone Joint Surg Br. 1995 May;77(3):377-83. PMID 7744919
- [Background] Matziolis G, Krocker D, Weiss U, Tohtz S, Perka C. A prospective, randomized study of computer-assisted and conventional total knee arthroplasty. Three-dimensional evaluation of implant alignment and rotation. J Bone Joint Surg Am. 2007 Feb;89(2):236-43. doi: 10.2106/JBJS.F.00386. PMID 17272435
- [Background] Siston RA, Patel JJ, Goodman SB, Delp SL, Giori NJ. The variability of femoral rotational alignment in total knee arthroplasty. J Bone Joint Surg Am. 2005 Oct;87(10):2276-80. doi: 10.2106/JBJS.D.02945. PMID 16203894
- [Background] Lutzner J, Krummenauer F, Wolf C, Gunther KP, Kirschner S. Computer-assisted and conventional total knee replacement: a comparative, prospective, randomised study with radiological and CT evaluation. J Bone Joint Surg Br. 2008 Aug;90(8):1039-44. doi: 10.1302/0301-620X.90B8.20553. PMID 18669959
- [Background] Weinrauch P, Myers N, Wilkinson M, Dodsworth J, Fitzpatrick P, Whitehouse S. Comparison of early postoperative rehabilitation outcome following total knee arthroplasty using different surgical approaches and instrumentation. J Orthop Surg (Hong Kong). 2006 Apr;14(1):47-52. doi: 10.1177/230949900601400111. PMID 16598087
- [Background] Kalairajah Y, Simpson D, Cossey AJ, Verrall GM, Spriggins AJ. Blood loss after total knee replacement: effects of computer-assisted surgery. J Bone Joint Surg Br. 2005 Nov;87(11):1480-2. doi: 10.1302/0301-620X.87B11.16474. PMID 16260662
- [Background] Victor J, Van Doninck D, Labey L, Innocenti B, Parizel PM, Bellemans J. How precise can bony landmarks be determined on a CT scan of the knee? Knee. 2009 Oct;16(5):358-65. doi: 10.1016/j.knee.2009.01.001. Epub 2009 Feb 5. PMID 19195896
- [Background] Henckel J, Richards R, Lozhkin K, Harris S, Rodriguez y Baena FM, Barrett AR, Cobb JP. Very low-dose computed tomography for planning and outcome measurement in knee replacement. The imperial knee protocol. J Bone Joint Surg Br. 2006 Nov;88(11):1513-8. doi: 10.1302/0301-620X.88B11.17986. PMID 17075100
- [Background] Kim S. Changes in surgical loads and economic burden of hip and knee replacements in the US: 1997-2004. Arthritis Rheum. 2008 Apr 15;59(4):481-8. doi: 10.1002/art.23525. PMID 18383407
- See also: Study description on website: Center for Implant and Radiostereometric Research Oslo - Oslo University Hospital — http://ous-research.no/cirro/?k=cirro%2FKnee+projects&aid=12521